CLINICAL TRIAL: NCT02284113
Title: A Post-Market, Multi-Center, Prospective, Double-Blind, Randomized, Controlled Study to Evaluate the Iovera° Device in Treating Pain Associated With Total Knee Arthroplasty
Brief Title: A Randomized, Study to Evaluate the Iovera° Device in Treating Pain Associated With Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MYO-1070
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Results first posted 2023-07-27 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Arthritis of the Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Treatment with focused cold therapy.
  Interventions: Device: iovera°
- Sham (Sham Comparator): Sham treatment with focused cold therapy device
  Interventions: Device: iovera° Sham

INTERVENTIONS:
Device: iovera° — Use of iovera° device to administer treatment Focused Cold Therapy
  Arms: Treatment
Device: iovera° Sham — iovera° device used for sham treatment
  Arms: Sham

SUMMARY:
This study will evaluate the iovera° device in treating pain associated with total knee arthroplasty (TKA). This study will also assess if overall pain medication is reduced following TKA and will investigate the relationship between patients treated with the iovera° device and length of hospital stay, pain, patient satisfaction and improved rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* 22 to 79 years of age
* Scheduled to undergo primary unilateral TKA under spinal anesthesia for primary diagnosis of osteoarthritis
* American Society of Anesthesiology (ASA) Physical Classification System classes I-III
* Anticipation of discharge to home after inpatient acute post-op phase (age, co-morbidities, home environment, and social support are in favor of discharge to home in the opinion of the Investigator)
* Subject is willing and able to give written informed consent.
* Subject is fluent in verbal and written English.
* Subject is willing and able to comply with study instructions and commit to all follow-up visits for the duration of the study.
* Subject is in good general health and free of any systemic disease state or physical condition that might impair evaluation or which in the Investigator's opinion, exposes the Subject to an unacceptable risk by study participation.

Exclusion Criteria:Exclusion Criteria

* Chronic opioid use (defined as daily or almost daily use of opioids for >3 months).
* Concurrent painful physical condition, surgery, or musculoskeletal disease that requires or may require analgesic treatment during study follow-up that is not strictly related to the target knee being treated with iovera°, which have the potential to confound the postoperative assessments (e.g., significant pain from other joints, chronic neuropathic pain, concurrent or planned contralateral TKA, concurrent foot, neck, spine, hip, or other musculoskeletal disease, arthritis, or planned surgery, etc.).
* Greater than 15° malalignment (varus or valgus) on pre-operative radiograph.
* Previous myoscience FCT™ treatment.
* Previous Partial or Total Knee Arthroplasty. Partial or Total Knee Arthroplasty of the contralateral knee is permitted if [surgery was completed at least twelve (12) months prior to screening].
* Body Mass Index ≥ 40
* Prior surgery in the treatment areas that may alter the anatomy of the infrapatellar branch of the saphenous nerve (ISN) or the anterior femoral cutaneous nerve (AFCN) or result in scar tissue in the treatment area.
* Any clotting disorder and/or use of an anticoagulant (e.g. warfarin, clopidogrel, etc.) within seven (7) days prior to administration of the device. Low dose aspirin (81mg or less daily) for cardiac prophylaxis allowed.
* Any local skin condition at the treatment sites that in the Investigator's opinion would adversely affect treatment or outcomes.
* Open and/or infected wound in the treatment areas.
* Allergy to lidocaine.
* History of cryoglobulinemia
* History of paroxysmal cold hemoglobinuria.
* History of cold urticaria.
* History of Raynaud's disease.
* History of opioid or alcohol abuse.
* Subject is pregnant or planning to become pregnant while enrolled in the study.
* Current enrollment in any investigational drug or device study or participation within 30 days prior to screening.
* Currently being treated for related knee injury under worker's compensation claim or equivalent (i.e. legal case).
* Any chronic medical condition that in the Investigator's opinion would prevent adequate participation.
* Any chronic medication use (prescription, over-the-counter, etc.) that in the Investigator's opinion would affect study participation or Subject safety.
* For any reason, in the opinion of the Investigator, the Subject may not be a suitable candidate for study participation (i.e., history of noncompliance, drug dependency, etc.).

Ages: 22 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-12; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California San Diego, San Diego, California
  - Colorado Orthopedic Consultants, P.C., Englewood, Colorado
  - Holy Cross Hospital Orthopedic Research Institute, Fort Lauderdale, Florida
  - Phoenix Clinical Research, LLC, Tamarac, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - LSUHSC - Department of Orthopaedics, New Orleans, Louisiana
  - Cleveland Clinic, Cleveland, Ohio
  - Rothman Institute, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Sham
Started | 74 | 76
Completed | 71 | 73
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 0
Not completed — non-compliance | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — not provided | 0 | 1
Not completed — surgery cancelled | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Sham | Total
Number analyzed (Participants) | 74 | 76 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (7.53) | 65.3 (9.33) | 65.3 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 45 | 83
  Male | 36 | 31 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 14 | 28
  White | 58 | 60 | 118
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 74 | 76 | 150
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.0 (4.61) | 30.6 (4.79) | 30.79 (4.69)

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Consumption of Opioids Total Daily Morphine Equivalent (TME) (mg/Day)
Description: The cumulative morphine equivalent was divided by the number of days to provide a Total Daily Morphine Equivalent (TME) for each Subject.
Time Frame: hospital discharge to 6 Weeks post-TKA surgery
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 69 | 71
mg/day | 23.9 (15.25) | 27.1 (20.87)

2. Secondary Outcome: Change in Pain From Baseline to Six Weeks
Description: The Numeric Rating Scale for Pain (NRS for Pain) is a measure of pain intensity which is assessed on a scale from 0 to 10 with 0 being no pain at all and 10 being the worst pain imaginable. The Subject provides a self-reported score based on their pain in the target knee at the time the questionnaire is administered (labeled 'now' in the tables below) as well as their pain in the past 7 days (labeled "past 7" in the tables below).
Time Frame: Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 73 | 75
score on a scale
  "Now" | -2.7 (2.96) | -3.6 (3.03)
  "Past 7 days" | -2.4 (3.01) | -2.9 (3.28)

3. Secondary Outcome: Change in WOMAC Scores at 6 Weeks After Surgery
Description: The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a tri-dimensional, disease-specific, Subject-reported outcome measure. It consists of 24 questions with 5 questions regarding pain, 2 questions regarding stiffness and 17 questions regarding function in Subjects with osteoarthritis of the hip and/or knee. Each question is answered on a scale of 0 (none)-10 (extreme). Higher scores are associated with worse outcomes.
Time Frame: Baseline to 6 weeks after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 73 | 75
score on a scale
  Pain | -13.1 (12.60) | -14.6 (13.18)
  Stiffness | -4.7 (5.29) | -5.5 (6.78)
  Physical Function | -49.4 (41.66) | -51.4 (44.56)

4. Secondary Outcome: Length of Hospital Stay
Time Frame: treatment to hospital discharge
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 71 | 73
Hours | 54.7 (27.34) | 52.6 (24.42)

5. Secondary Outcome: Change in Active Range of Motion From Baseline to 2 Weeks After Surgery
Description: Range of motion measures the physical function of the replaced knee during active flexion at the specified timepoints.
Time Frame: baseline to 2 weeks after surgery
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 73 | 73
Degrees | -10.1 (19.51) | -11.8 (15.56)

6. Secondary Outcome: 40 Meter Walk Test
Description: The 40 Meter Walk Test measured the average speed in meters per second a Subject could walk 40 meters.
Time Frame: Baseline, 2,4,6,12 weeks
Population: The variation in number analyzed is due to the actual number of participants with data collected at specific timepoint
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 74 | 76
meters per second
  Baseline | 1 (0.41) | 1 (0.42)
  2 weeks: number analyzed (Participants) | 69 | 71
  2 weeks | 0.8 (.34) | 0.8 (.31)
  4 weeks: number analyzed (Participants) | 66 | 70
  4 weeks | 0.9 (0.31) | 0.9 (0.34)
  6 weeks: number analyzed (Participants) | 73 | 73
  6 weeks | 1.0 (0.34) | 1.0 (0.38)
  12 weeks: number analyzed (Participants) | 73 | 72
  12 weeks | 1.1 (0.35) | 1.1 (0.36)

7. Secondary Outcome: 30 Second Chair Test
Description: The 30 Second Chair Test evaluates physical function during recovery by measuring the number of times a subject could go from seated in a chair to standing over the course of 30 seconds.
Time Frame: Baseline, 2,4,6,12 weeks after surgery
Population: The variation in number analyzed is due to the actual number of participants with data collected at specific timepoint
Measure: Mean (Standard Deviation); unit: number of repetitions
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 74 | 76
number of repetitions
  Baseline | 8.2 (3.38) | 8.6 (4.34)
  2 weeks: number analyzed (Participants) | 69 | 71
  2 weeks | 6.9 (3.26) | 7.5 (3.07)
  4 weeks: number analyzed (Participants) | 66 | 70
  4 weeks | 9.6 (3.81) | 9.5 (3.81)
  6 weeks: number analyzed (Participants) | 73 | 73
  6 weeks | 12.4 (13.75) | 11.1 (3.93)
  12 weeks: number analyzed (Participants) | 73 | 72
  12 weeks | 12.1 (4.31) | 13.0 (4.11)

8. Secondary Outcome: Change 36-Item Short Form Health Survey (SF-36) From Baseline to 6 Weeks
Description: The 36-question survey captures the Subject's perception of their general health by sorting them into multi-item scales that assess eight health concepts rather than a single total score. The survey used ten components to assess the health concepts: Physical, Mental, Physical Functioning, Role- Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role Emotional, and Health Transition. Subject responses to the SF-36 survey were recorded. Scores can range from 0 to 100. Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales.
Time Frame: Baseline to Week 6
Population: The variation in number analyzed is due to the actual number of participants with data collected at specific timepoint
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 73 | 75
change in score on a scale
  Physical Component | 3.8 (7.70) | 6.3 (9.58)
  Mental Component: number analyzed (Participants) | 72 | 75
  Mental Component | 0.7 (10.73) | 0.3 (10.61)
  Physical Functioning | 13.6 (23.83) | 16.7 (28.49)
  Role-Physical Component: number analyzed (Participants) | 72 | 75
  Role-Physical Component | 4.3 (31.83) | 17.8 (33.67)
  Bodily Pain Component | 13.2 (23.07) | 16.9 (26.66)
  General Health Component | 1.7 (12.18) | 1.5 (14.17)
  Vitality Component | 3.2 (20.15) | 4.2 (17.78)
  Social Functioning Component | 4.3 (30.56) | 4.5 (27.54)
  Role Emotional: number analyzed (Participants) | 72 | 75
  Role Emotional | 0.7 (32.61) | 7.4 (34.62)
  Health Transition Component | -0.5 (1.13) | -0.07 (1.12)

9. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS) From Baseline to Week 6
Description: 8 domains assessing physical, mental and social health while also covering important areas of self-reported health: pain, fatigue, depression, anxiety, sleep, and physical function. A high PROMIS domain sub-score indicates more of that concept being measured. PROMIS scores have a mean of 50 and standard deviation (SD) of 10 in a referent population. The referent population is usually the US General Population. lower scores are less favorable, and higher scores are more favorable.
Time Frame: Baseline to 6 weeks after surgery
Population: The variation in number analyzed is due to the actual number of participants with data collected at specific timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Sham
Number analyzed (Participants) | 73 | 75
score on a scale
  Physical Function: number analyzed (Participants) | 72 | 75
  Physical Function | -2.3 (4.36) | -2.6 (4.50)
  Anxiety | -1.0 (3.17) | -1.2 (2.94)
  Depression | -0.3 (2.47) | 0.1 (2.85)
  Fatigue | 9.6 (3.74) | 8.7 (3.79)
  Sleep Disturbance: number analyzed (Participants) | 73 | 74
  Sleep Disturbance | 0.1 (1.83) | 0.22 (1.98)
  Ability to Participate in Social Roles and Activities: number analyzed (Participants) | 73 | 74
  Ability to Participate in Social Roles and Activities | -0.3 (4.48) | -0.6 (3.83)
  Pain Interference: number analyzed (Participants) | 72 | 75
  Pain Interference | -2.5 (4.55) | -2.8 (4.56)
  Pain Intensity | -2.6 (2.8) | -3.3 (2.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Visit 2/Treatment through Visit 7/12 weeks post-op
Arm/Group | Treatment | Sham
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/76
Serious Adverse Events (participants affected / at risk) | 5/74 | 5/76
Other Adverse Events (participants affected / at risk) | 24/74 | 24/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=74) | Sham (N=76)
Staphylococcal infection Left Hand (Infections and infestations) | 0 (0) | 1 (1)
Incision site Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Elevated white blood count (Investigations) | 1 (1) | 0 (0)
Acute Kidney Injury CKD Stage 3 (Renal and urinary disorders) | 0 (0) | 1 (1)
Chest pain, left arm numbness (General disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Infection Left knee-Post TKA (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess left buttocks (Infections and infestations) | 0 (0) | 1 (1)
Left Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=74) | Sham (N=76)
Bursitis Knee (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
knee arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Cellulitis around incision (Infections and infestations) | 0 (0) | 3 (3)
peripheral edema of lower leg (General disorders) | 2 (3) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hemarthrosis acute (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2015-05-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT02284113/Prot_000.pdf